CLINICAL TRIAL: NCT05102682
Title: Rex Robot Assisted Rehabilitation Exercise to Enhance Balance, Mobility and Upper Limb Function in People With Multiple Sclerosis
Brief Title: Robotics for Mobility Rehabilitation in MS
Acronym: RAPPERIII
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: REC reference: 16/EE/0553
Record Dates: First submitted 2021-10-25; First posted 2021-11-01 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis; MS
Keywords: Neurorehabilitation; Feasibility; exoskeleton
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Prospective, open label, single arm, non-randomized, non-comparative feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance rehabilitation exercise (Experimental): Balance rehabilitation exercise program using exoskeleton device
  Interventions: Other: Balance exercise program using exoskeleton device

INTERVENTIONS:
Other: Balance exercise program using exoskeleton device — Exercise program focused on strengthening core body muscles and balance supported by Rex exoskeleton device

SUMMARY:
Title Prospective, open label, single arm, non-randomized, non-comparative feasibility study of Rex robot assisted rehabilitation exercise to enhance balance, mobility and upper limb function in people with Multiple Sclerosis "RAPPER III - MS Objective The objective of this study is to evaluate the feasibility and safety of the REX Robot when used for rehabilitation with people who have moderate to severe mobility restrictions due to MS. A secondary objective of the study is to explore the acceptability of the device to people with MS and its impact on impairments and functions commonly affected by MS.

Study Sponsor Rex Bionics, Plc. Study Device REX Robotic powered exercise system Primary Endpoint • Completion of a transfer, stand, balance and walk rehabilitation session.

* Unexpected Serious Adverse Events Secondary Endpoints
* Completion of a transfer, stand, balance and walk rehabilitation program over Six-weeks
* The Number of approached, screened, and eligible potential participants. Reasons for Ineligibility. (See 'RAPPER III- MS 007 Screening Loss Analysis REV 0 FINAL')
* Functional Ambulation Classification (FAC) 1
* Activities-specific Balance Confidence (ABC) Scale 2
* Modified Falls Efficacy Scale (MFES) 3, 4,
* Multiple Sclerosis Walking scale (MSWS-12) 5
* Multiple Sclerosis Impact scale (MSIS-29) 6
* ARMA (arm activity measure) 7
* Berg Balance Scale 8
* Timed unsupported steady stand (TUSS) 9
* Pain scale questionnaire (Visual Analog Score VAS) 10
* Modified Ashworth Score 11
* Spasticity Impact Scale 12
* Epworth Sleepiness Scale (ESS) questionnaire 13
* EQ-5D Health State Questionnaire 14

Questionnaires may be administered in person, by phone, email or in the post.

DETAILED DESCRIPTION:
Participant Information Sheet Study title: Rex robot Assisted rehabilitation exercise to enhance balance, mobility and uPPER limb function in people with Multiple Sclerosis "RAPPER III - MS"

Rex Bionics are now enrolling for RAPPER III, a 10 patient trial at East Kent University Hospital foundation Trust.

The study will take place at the following address:

School Of Engineering and Arts, Jennison Building, University of Kent, Canterbury CT2 7NT We would like to invite you to take part in our research study. Before you decide we would like you to understand why the research is being done and what it would involve for you. One of our team will go through the information sheet with you and answer any questions you have.

The objective of this feasibility study is to evaluate the overall device safety when used in a Clinical Rehabilitation Centre under the supervision of a physician and/or qualified rehabilitation specialist. The trial can be completed by patients over 6 sessions, each a week apart. The study will consist of walking in REX Bionics powered exercise device and completing a variety of therapy exercises the assistance of REX trained therapists. You will be asked to complete some questionnaires and other tests before the first session, after the 3rd session and finally after your 6th session.

This document is broken into 2 parts Part 1 - tells you the purpose of this study and what to expect if you take part.

Part 2 - gives you more detailed information about the conduct of the study. Part 1 What is the purpose of this study?

i) To assess the feasibility and safety of undertaking a neuro-rehabilitation exercise program using a Rex robotic device within a controlled clinical environment (ease of use for both user and therapist ii) Investigate the potential to improve balance and walking using Rex for people with MS iii) Investigate the potential health benefits of this Rex Rehabilitation program iv) Ascertain whether there might be a measurable impact on upper limb functional abilities

Why have I been invited? You have been asked to participate in this study because you have a diagnosis of multiple sclerosis that fits the inclusion criteria of this study. There will be a number of assessments prior to trialling the device to ensure you fit the criteria to safely use REX. This is for your own safety.

Do I have to take part? It is up to you to decide to join the study. We will describe the study and go through the information sheet. If you agree to take part, we will then ask you sign a consent form. You are free to withdraw at any time, without giving a reason. This would not affect the standard of care you receive. We are planning to enrol 10 people for this study.

What will happen to me if I take part? Study Schedule You will be asked to come to the rehab clinic for 6 sessions. The timing of these sessions vary and more detail is given below. Each session will be a week apart. Please ensure you wear supportive fitting laced shoes, a pair of comfortable sporting trousers/track suit bottoms and a light T-Shirt or Similar. If you have issues with the support structures of your feet you should consider using orthotics to offer added support. Please raise any concerns you have with your therapist conducting the research so further information can be provided to you.

* Enrolment - You will be asked some screening questions prior being enrolled in the study. If you are enrolled, you will be asked to complete 13 outcome measures (tests/questionnaires) in session 1, 4 questionnaires 2 days after session 3 and finally all 13 outcome measures (tests/questionnaires) in session 6. (approximately 90 minutes)
* Session 1 - you will be asked to come into the clinic to complete a number of tasks. (approximately 150 minutes)

Task 1: baseline medical assessment and giving informed consent:

A medical examination will take place along with a discussion around your current medical conditions and previous medical conditions to determine if you are safe to use REX.

You will be given a patient information sheet and ask to give consent if you would like to be included in the study. You can withdraw at any time and do not have to give consent if you do not choose to.

Task 2: Assessment against inclusion criteria:

You will be assessed against a number of different inclusion and exclusion criteria to determine whether you are appropriate for the study

Task 3: completion of pre-treatment outcome measures and questionnaires:

You will be asked to complete a number of scales and questionnaires. These will be repeated at the end of the study (during sessions 6). If you have any questions about any of these you should ask the investigator and the investigator will provide you with enough time and space to discuss everything. The outcome measures are listed below.

* Activities-specific Balance Confidence (ABC) Scale
* Modified Falls Efficacy Scale (MFES)
* Multiple Sclerosis Walking scale (MSWS-12)
* Multiple Sclerosis Impact scale (MSIS-29)
* ARMA (arm activity measure)
* Berg Balance Scale
* Video of sit to stand and stand to sit (recorded twice )
* Video of walking - timed up and go (3 metres )
* Pain scale questionnaire (Visual Analog Score VAS)
* Modified Ashworth Score
* Epworth Sleepiness Scale (ESS) questionnaire
* EQ-5D Health State Questionnaire Task 4: Measurements, fitment and mobilizing A number of measurements will be taken to ensure you can safely use and fit the device Once these have been taken you will be asked to transfer into the device. This will be timed.

On completion of a safe transfer you will be asked to stand up in Rex and walk 3 m, turn around and come back again, then sit back down on the chair. This will be timed.

Task 5: Exercise prescription The investigator will work with you to determine an appropriate amount of weights/resistance that should be used for your treatment programs in the subsequent session.

Session 2: Completion of a prescribed exercise program. (approximately 45 minutes) Task 1: You will be asked to complete a set number of exercises that should last approximately 45 minutes.

Session 3: completion of a prescribed exercise program. (approximately 45 minutes) Task

Task 2: You will be asked to complete 3 questionnaires 2 days (plus or minus one day for flexibility with your schedule) after your exercise program. These will be completed over the phone with the investigator conducting the study. You will be given an envelope with all the questionnaires in so you have a point of reference. These questionnaires will be:

* Pain scale questionnaire (Visual Analog Score VAS)
* Epworth Sleepiness Scale (ESS) questionnaire You will also be assessed for your level of spasticity using the Modified Ashworth Score
* Session 4: Completion of a prescribed exercise program. (approximately 60 minutes) Task 1: you will be asked to complete a set number of exercises as you did in the previous sessions
* Session 5: completion of a prescribed exercise program. (approximately 60 minutes) Task 1: you will be asked to complete a set number of exercises as you did in your previous sessions Task 2: You will be asked to complete a timed transfer to see if it has got any quicker since your first session.
* Session 6: Completion of follow up outcome measures and questionnaires. (approximately 90 minutes) Task 1: You will be asked to complete all the same scales and questionnaires you completed in session 1 to see if there has been any improvement.

If you are unable to make the appointed visits in the time frame above, you will need to notify your physician or rehabilitation therapist.

What are the possible disadvantages and risk of taking part?

* Accidental injury due to falling
* Skin issues such as bruising and redness
* Complications with you blood pressure
* Risks of breaks or fractures through falling
* Hip subluxation/instability
* Risk of Autonomic Dysreflexia with spinal cord injuries of T6 and above
* Risk of unintended bowel movement due to movement in REX

What are the possible benefits of taking part? You might not get benefits from the study, however a greater understanding of whether the REX System can be used to rehabilitate patients with a similar condition will be gained from your participation in this study. This information may contribute to the development of new treatments for persons with Multiple Sclerosis.

What if there is a problem? Any complaint about the way you have been dealt with during the study or any possible harm you might suffer will be addressed. The detailed information on this will be provided in part 2.

Will the taking part in the study be kept confidential? Yes. The records obtained while you are in this study as well as related health records will be strictly confidential at all times under the provisions of the 1998 Data Protection Act, to enable analysis of the study results. With your permission, you're GP and other doctors who may be treating you will be notified that you are taking part in this study. Further details are included in part 2.

In case of an adverse event your GP will be contacted and informed.

If the information in part 1 has interested you and you are considering participation, please read the additional information in part 2 before making any decision.

Part 2:

What if relevant new information becomes available? Sometimes we get new information about the treatments being studied. If this happens, your local research team will tell you and discuss whether you should continue in the study. You can withdraw from the study at any time.

What will happen if I don't want to carry on with the study? Taking part in this research study is voluntary. You may decide to stop at any time. You should tell the researcher if you decide to stop, this would not affect the standard of care you receive.

In addition, the researchers, Rex Bionics, or your hospital or clinic may stop you from taking part in this study at any time:

* if it is in your best clinical interest,
* if you do not follow the study procedures,
* If the study is stopped.

What if there is a problem? If you have a concern about any aspect of this study, you should ask to speak to the researchers who will do their best to answer your questions. If you remain unhappy and wish to complain formally, you can do this by contacting Mohammed Sakel the Chief Investigator for NHS sites at msakel@nhs.net. Alternatively you can contact Mathew Pepper at matthew.pepper@nhs.net or Karen Saunders at karensaunders1@hotmail.com

Will You Be Paid For Participating In This Research Study?

No. But you will be provided with a 50 pound gift voucher for M&S. Free parking will also be provided when you attend at the clinic.

What Happens if You Are Injured Or Ill In The Course of this Study?

Where to get help:

If you think you have suffered a research-related injury, you should promptly notify the Principal Investigator listed in the Contact Information at the end of this form. The Hospital or Clinic will offer care for research-related injuries, including first aid, emergency treatment and follow-up care as needed.

Who will pay for the treatment of research related injuries?

If you have side effects from the study treatment, you need to report them to the researcher and your regular physician, and you will be treated as needed. If you have injuries directly resulting from the application of the study device or procedures, whether at your health care provider or another institution, the Sponsor, Rex Bionics will pay for appropriate medical treatment beyond that covered by your health insurance or other third party or government programs, at no cost to you. Your study doctor can help you obtain this reimbursement. Sponsor will not be responsible for deductibles and co-pays.

Authorization to Use and Disclose Protected Health Information Your privacy is important to us, and we want to protect it as much as possible. By signing the consent form, you authorize the Hospital or Clinic and the investigators to use and disclose any information created or collected in the course of your participation in this research protocol. This information might be in different places, including your original medical record, but we will only disclose information that is related to this research protocol for the purposes listed below.

This information will be given out for the proper monitoring of the study, checking the accuracy of study data, analysing the study data, and other purposes necessary for the proper conduct and reporting of this study. If some of the information is reported in published medical journals or scientific discussions, it will be done in a way that does not directly identify you.

This information may be given to other researchers in this study, including those at other institutions, representatives of the company sponsoring the study, including representatives in your country or other countries, or private, state or federal government parties or regulatory authorities in your country and other countries responsible for overseeing this research. These may include the US Food and Drug Administration, the Office for Human Research Protections, or other offices in your country within the Department of Health

Information Disclosed to Study Sponsor The study data sent by the study doctor to the sponsor does not include your name, address, ID number, or other information that directly identifies you. Instead, the study doctor assigns a code number to the study data and may use your initials. Some study data sent to the sponsor may contain information that could be used (perhaps in combination with other information) to identify you (e.g. date of birth). If you have questions about the specific health information that will be sent to the sponsor, you should ask the study doctor.

This authorization lasts until the end of the study. The study does not end until all data has been collected, checked (or audited) and analysed. Sometimes this can be years after your study visits have ended. For example, this could happen if the results of the study are filed with a regulatory agency like the local regulatory authorities or US Food and Drug Administration.

You may stop this authorization at any time by writing to the following address:

Mohamed Sakel Director/Consultant Neurorehabilitation Physician East Kent University NHS FT hospitals Canterbury UK CT13NG

If you stop authorization, the hospital or Rehab centre may continue to use your information already collected as part of this study, but will not collect any new information.

If you do not sign this authorization, or later stop authorization, you may not be able to participate in the study.

What Will Happen to Your Data after?

Your data will be used as described for this study. When the study is done, they may be used for the purpose of publication, your name or identity will NEVER be revealed.

Who Can Answer Your Questions?

You can call the

Principal Investigator: Mohamed Sakel

Study Coordinator:

Phone: 00447500817652

ELIGIBILITY:
Inclusion Criteria:

Have a confirmed diagnosis of MS by a Consultant Neurologist as per Mc Donald Criteria. Have moderate to severe mobility restriction as defined by an Extended Disability Status Scale (EDSS) score of between 6 to 7.5 (inclusive). Meet the anthropometric requirements of the REX device (See 'RAPPER IIIMS 014 TF-04 v 3.0 REX Clinical Assessment Guide A4' for details of weight, height, size and range of motion requirements) Offer written informed consent to take part in the study

Exclusion Criteria:

a history of osteoporosis or osteoporosis related bone fractures. skin integrity issues that could be adversely affected by the REX device severe hypertonia (spasticity) as indicated by a score equal to or greater than 4 on the modified Ashworth scale on any muscle in their lower limbs. a behavioural, cognitive or communication impairment which could interfere with the ability to participate in a rehabilitation programme, as noted during screening (e.g., agitation, inability to follow two step commands) Are unable or unwilling to provide informed consent Are considered medically unsuitable for rehabilitation in the opinion of the screening medical specialist a known allergy (skin contact) to materials used in Rex Are pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
Completion and time taken for participant transfer into Rex device | First trial session
  Timed transfer into device (seconds)
Completion of sit to stand in Rex device by participant | First trial session
  Participant inside Rex device with device switched on moves from sit to stand with supervision of therapist
Completion of 1 timed 3 metre walk in device (Timed Up & Go Test) | First trial session
  Participant completes timed walk as above with assistance and guidance from therapist
Completion of trial sessions | 6 sessions in total
  Completion of all 6 trial sessions noted and recorded in records

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Dr Sakel, MBBS, Principal Investigator — East Kent Hospitals University NHS Foundation Trust
Locations (1):
- East Kent Hospitals University NHS Trust, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No